CLINICAL TRIAL: NCT00487422
Title: A Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy, Safety and Quality-of-Life of R108512 Tablets in Elderly Subjects With Chronic Constipation
Brief Title: Efficacy and Safety Study of Prucalopride for the Treatment of Elderly Patients With Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRU-INT-12
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2007-06

CONDITIONS: Constipation
Keywords: constipation; prucalopride; QOL; SCBM; PAC-SYM
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Prucalopride
  Interventions: Drug: prucalopride
- 2 (Active Comparator): Prucalopride
  Interventions: Drug: Prucalopride
- 3 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: prucalopride — 2 mg o.d.
  Other Names: Resolor
  Arms: 1
Drug: Prucalopride — 4 mg o.d.
  Other Names: Resolor
  Arms: 2
Other: Placebo — o.d.
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether prucalopride is safe and effective in the treatment of chronic constipation in elderly patients.

Hypothesis:

Prucalopride 2 mg and 4 mg given once daily for 12 weeks is superior to placebo for the treatment of patients with chronic constipation and is well tolerated in those patients

DETAILED DESCRIPTION:
This is a multicentre, randomised, Phase III trial with a parallel-group design, consisting of a 2 week drug-free run-in period, followed by a 4-week, double-blind, placebo-controlled treatment period.

During the run-in period, the subject's bowel habit will be documented and the existence of constipation confirmed. At the start of this period, all existing laxative medication will be withdrawn and subjects will be instructed not to change their diet or lifestyle during the trial.

Subjects will be allowed to take a laxative (Dulcolax®) as a rescue medication throughout the trial, but only if they have not had a bowel movement for three or more consecutive days. Subjects will enter the double-blind period if constipation is shown to be present during the run-in period. Patients will be randomly allocated to one of the 4 treatment arms: 1 mg, 2 mg, 4 mg of R108512 or placebo, with a 25% chance to each treatment group.

During the double-blind period, subjects will be treated for 4 weeks with either 1 mg, 2 mg or 4 mg R108512 or placebo, given once daily before breakfast.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects of 65 or over 65 years of age.
2. History of constipation; the subject reports, on average, two or fewer spontaneous bowel movements per week that result in a feeling of complete evacuation and one or more of the following for at least 6 months before the selection visit:

   1. very hard (little balls) and/or hard stools at least a quarter of the stools
   2. sensation of incomplete evacuation following at least a quarter of the stools
   3. straining at defecation at least a quarter of the stools. The above criteria are only applicable for spontaneous bowel movements, i.e., not preceded within a period of 24 hours by the intake of a laxative agent or by the use of an enema.

Subjects who never have spontaneous bowel movements are considered to be constipated and are eligible for the trial.

Exclusion Criteria:

1. Subjects in whom constipation is thought to be drug-induced, or subjects using any disallowed medication.
2. Subjects suffering from endocrine disorders, metabolic disorders or neurologic disorders.
3. Subjects with the main complaint of abdominal pain.
4. Subjects with a known megacolon/megarectum or a diagnosis of pseudo-obstruction.
5. Constipation as a result of surgery.
6. Known or suspected organic disorders of the large bowel, i.e. obstruction, carcinoma, or inflammatory bowel disease.
7. Malignancies or AIDS.
8. Known serious illnesses: clinically significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, psychiatric or metabolic disturbances. Patients with known diverticulosis may be included.
9. Subjects with a serum creatinine concentration > 2 mg/dL (> 180 micromol/L).
10. Subjects with clinically significant abnormalities of haematology, urinalysis, or blood chemistry.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 303 (Actual)
Dates: Start 1998-10; Primary Completion 1999-09 (Actual); Study Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an average of 3 or more SCBM per week | 12 weeks

SECONDARY OUTCOMES:
Secondary efficacy variables: 1)Symptom variables 2)QOL variables | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Demschik, M.D., Principal Investigator — Geriatriezentrum am Wienerwald

REFERENCES:
- [Derived] Muller-Lissner S, Rykx A, Kerstens R, Vandeplassche L. A double-blind, placebo-controlled study of prucalopride in elderly patients with chronic constipation. Neurogastroenterol Motil. 2010 Sep;22(9):991-8, e255. doi: 10.1111/j.1365-2982.2010.01533.x. Epub 2010 Jun 7. PMID 20529205